CLINICAL TRIAL: NCT02603198
Title: 2%-Mepivacaine With Two Different Vasoconstrictors; 1:20.000 Levonordefrin or 1:100.000 Epinephrin for Local Anesthesia in Third Molar Surgery: A Comparative Randomized Clinical Trial
Brief Title: 2%-Mepivacaine With Two Different Vasoconstrictors Solutions in Third Molar Surgery a Comparative Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Maria Cristina Zindel Deboni, Associate Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 34147114500000068
Record Dates: First submitted 2015-11-08; First posted 2015-11-11 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Pain; Trismus; Edema
Keywords: third molar; tooth extraction; impacted tooth
MeSH Terms: conditions — Pain; Trismus; Edema; Tooth, Impacted | interventions — Anesthesia, Local

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- mepivacaine chloridrato epinephrine (Active Comparator): Side of operation that is going to receive anesthesia with 2% mepivacaine chloridrato with 1:100.000 epinephrine, maximum of 4 cartridges
  Interventions: Drug: mepivacaine chloridrato epinephrine
- mepivacaine chloridrato levonordefrin (Active Comparator): Side of operation that is going to receive anesthesia with 2% mepivacaine chloridrato with 1:20.000 levonordefrin, maximum of 4 cartridges
  Interventions: Drug: mepivacaine chloridrato levonordefrin

INTERVENTIONS:
Drug: mepivacaine chloridrato epinephrine — local anesthesia for tooth removal
  Other Names: local anesthesia
  Arms: mepivacaine chloridrato epinephrine
Drug: mepivacaine chloridrato levonordefrin — local anesthesia for tooth removal
  Other Names: local anesthesia
  Arms: mepivacaine chloridrato levonordefrin

SUMMARY:
Dental treatments, particularly third molars extraction, can become extremely uncomfortable and painful. They are associated to anxiety, fear and many other unpleasant sensations. During surgery, patients can present cardiorespiratory repercussions of these sensations. This fact generally justifies the employment of methods of monitoring and appliance of safer therapeutic alternatives. Local anesthetics are the most frequently drugs used in dentistry. Vasoconstrictors, particularly epinephrine, are important components of anesthetic solutions to increased time for anesthetic absorption and consequently increasing the duration of anesthesia. The use of smaller amounts of anesthetic solution can reduce the risk of systemic toxicity, however decrease the total surgical time. It is well known that the amount of epinephrine injected into patients during anesthetic procedures can produce adverse hemodynamic effects. Levonordefrin was adding to dental cartridges promising to reduce cardiac stimulation due it less β activity, and maintain the same clinical and systemic effects. But some studies for maxillary or intraosseous infiltrations showed no difference in heart rate and any anesthetic success over epinephrine. Thus, this study aims to compare the clinical efficacy and safety of anesthetic mepivacaine 2% with epinephrine 1:100,000 or 1:20,000 levonordefrin employing a clinical trial model of third molars extractions in healthy adults.

DETAILED DESCRIPTION:
30 healthy patients, both gender between 18 and 40 years-of-age with the necessity of bilateral third molar removal with similar surgical difficulty will be recruited from a Dental Public University Clinic. Inclusion criteria includes: non-smoking participants, minimum of 50 Kg of weight. After clinical and radiographic examination, they will be randomized accordingly to the side to be operated in two groups: MEPI-LEVO and MEPI-EPI. There will be a memory-washout of 15days between surgeries. In the MEPI-LEVO group, the patient will receive local anesthesia employing 2% chloridrato mepivacaine with 1:20.000 levonordefrin at a maximum of four cartridges of anesthesia. The other side will receive 2%chloridrato mepivacaine with 1:100.000 epinephrine in the same maximum amount. The surgery in both groups will follow strictly patterns of minimum surgical trauma and high cautious antiseptic conditions. The same surgeon will do the tooth extractions but the anesthesia will be done by another oral surgeon in order to blind the type of anesthetic solution from the operator (type of vasoconstrictor used). The amount of bleeding will be quantified just immediately after suture by a blinded observer that will record in a visual analogical scale between 0 and 10 points, where 0 correspond to absence of bleeding and 10 to excessive bleeding.

Blood pressure and heart rate will be accessed in five different moments:

1. 20minutes before surgical procedure with patients in awaiting room;
2. 5 minutes before procedure with patient seated in dental chair;
3. 5 minutes after anesthesia procedure;
4. during osteotomy/tooth sectioning and
5. after 10 minutes of suturing.

Patients after surgery will receive a diary to record the time when anesthesia sensation had ended, the amount of analgesics they had consumed and the level of pain in a visual analogic scale. The data will be submitted to statistical analysis with p<0.05 of significance.

ELIGIBILITY:
Inclusion Criteria:

* minimum body weight of 50Kg, necessity of bilateral impacted third molar removal

Exclusion Criteria:

-

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-08; Primary Completion 2015-06 (Actual); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Change in Blood pressure values | 20 minutes pre-operatory, 5 minutes before surgery, 5 minutes after anesthesia, 10 minutes after suture
  assessment of blood pressure values (systolic and diastolic)) in mmHg by a pulse electronic device

SECONDARY OUTCOMES:
Change in Heart Rate values | 20 minutes pre-operatory, 5 minutes before surgery, 5 minutes after anesthesia, 10 minutes after suture
  assessment of Heart Rate in bpm (beats per minute) by a pulse electronic device
Bleeding | after 1 hour postoperatively
  Assessment by a visual analogical scale - blinded observer record
Pain | 6, 8,24 and 48 hours after suture
  assessment by visual Analogical Scale - Patient diary

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo Minharro Cechetti, PhD, Principal Investigator — Post - Doctorate
Locations (1):
- Maria Cristina Zindel Deboni, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ezmek B, Arslan A, Delilbasi C, Sencift K. Comparison of hemodynamic effects of lidocaine, prilocaine and mepivacaine solutions without vasoconstrictor in hypertensive patients. J Appl Oral Sci. 2010 Jul-Aug;18(4):354-9. doi: 10.1590/s1678-77572010000400006. PMID 20835569
- [Background] Hersh EV, Giannakopoulos H. Beta-adrenergic blocking agents and dental vasoconstrictors. Dent Clin North Am. 2010 Oct;54(4):687-96. doi: 10.1016/j.cden.2010.06.009. PMID 20831932
- [Background] Serrera Figallo MA, Velazquez Cayon RT, Torres Lagares D, Corcuera Flores JR, Machuca Portillo G. Use of anesthetics associated to vasoconstrictors for dentistry in patients with cardiopathies. Review of the literature published in the last decade. J Clin Exp Dent. 2012 Apr 1;4(2):e107-11. doi: 10.4317/jced.50590. eCollection 2012 Apr. PMID 24558534
- [Background] Pellicer-Chover H, Cervera-Ballester J, Sanchis-Bielsa JM, Penarrocha-Diago MA, Penarrocha-Diago M, Garcia-Mira B. Comparative split-mouth study of the anesthetic efficacy of 4% articaine versus 0.5% bupivacaine in impacted mandibular third molar extraction. J Clin Exp Dent. 2013 Apr 1;5(2):e66-71. doi: 10.4317/jced.50869. eCollection 2013 Apr 1. PMID 24455059
- [Background] Torres-Lagares D, Serrera-Figallo MA, Machuca-Portillo G, Corcuera-Flores JR, Machuca-Portillo C, Castillo-Oyague R, Gutierrez-Perez JL. Cardiovascular effect of dental anesthesia with articaine (40 mg with epinefrine 0,5 mg % and 40 mg with epinefrine 1 mg%) versus mepivacaine (30 mg and 20 mg with epinefrine 1 mg%) in medically compromised cardiac patients: a cross-over, randomized, single blinded study. Med Oral Patol Oral Cir Bucal. 2012 Jul 1;17(4):e655-60. doi: 10.4317/medoral.17892. PMID 22322521
- [Background] Lawaty I, Drum M, Reader A, Nusstein J. A prospective, randomized, double-blind comparison of 2% mepivacaine with 1 : 20,000 levonordefrin versus 2% lidocaine with 1 : 100,000 epinephrine for maxillary infiltrations. Anesth Prog. 2010 Winter;57(4):139-44. doi: 10.2344/0003-3006-57.4.139. PMID 21174567